CLINICAL TRIAL: NCT06991036
Title: Validation of Plant-Based Vegan Meal for Gastric Emptying Testing in 10 Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 24-008112
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gastric Emptying; Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard egg meal then vegan meal (Experimental): At first visit, gastric emptying test will be performed on subjects after consuming the standard egg meal consisting of two large whole, scrambled chicken eggs, one slice of wheat bread, and one glass (around 236 mL) of skim milk and provided approximately 320 kcal and 30% fat.
  Approximately 1 week later, the gastric emptying test will be performed again after subjects consume the vegan breakfast meal consisting of around 4 fl oz of JUST Egg® (a plant-based egg substitute) which is primarily made from mung beans, two slices of gluten-free multigrain bread, 4 fl oz of orange juice, and ½ a cup of water.
  Interventions: Other: Gastric emptying test
- Vegan meal then standard egg meal (Experimental): At first visit, gastric emptying test will be performed on subjects after consuming the vegan breakfast meal consisting of around 4 fl oz of JUST Egg® (a plant-based egg substitute) which is primarily made from mung beans, two slices of gluten-free multigrain bread, 4 fl oz of orange juice, and ½ a cup of water.
  Approximately 1 week later, the gastric emptying test will be performed again after subjects consume the standard egg meal consisting of two large whole, scrambled chicken eggs, one slice of wheat bread, and one glass (around 236 mL) of skim milk and provided approximately 320 kcal and 30% fat.
  Interventions: Other: Gastric emptying test

INTERVENTIONS:
Other: Gastric emptying test — After the radiolabeled breakfast meal is ingested, the participant is positioned upright between the two detectors of the Brightview system (Phillips Medical Systems, Cleveland, OH). Detector height is adjusted to include esophageal uptake, the stomach, and the small bowel. Anterior and posterior static images are acquired at 2 minutes per image using a 256 x 256 word mode matrix. Anterior and posterior images are again acquired at 1 and 2 hours post-ingestion of the radiolabeled breakfast meal.
  The participant is then given the designated 'push' meal after completion of the 2-hour images. At 4 hours post-ingestion, images are acquired in the same manner as at previous time points.

SUMMARY:
The purpose of this research study is to compare the stomach emptying function using a current standard meal which includes eggs and our new vegan meal alternatives for patients who are not able to eat eggs.

DETAILED DESCRIPTION:
10 healthy participants underwent randomized crossover (with concealed allocation) GE scintigraphy with standard and vegan meals, spaced ≥3 days apart to measure GE% at 2h, 4h, and GE T1/2. Group comparisons and variance analysis included Rank Sum tests and Bland-Altman plots.

ELIGIBILITY:
Inclusion Criteria:

* No history of diabetes
* Not on medications that affect gastric emptying without diagnosis of active gastrointestinal disease
* No history of prior gastrointestinal surgery that would interfere with testing
* No recent (within last 10 years) gastritis, gastrointestinal infections, COVID-19 (within last 2 years), H pylori, peptic ulcer disease
* Not pregnant,
* Not actively breast-feeding
* No history of stomach cancers
* No history of neurodegenerative disorder
* Able to sign informed consent and take part in study
* BMI <35

Exclusion Criteria:

* History of diabetes
* Taking medications that affect gastric emptying (e.g., GLP-1 agonists, opioids, calcium channel blockers, pramlintide, tricyclic antidepressants, buspirone)
* Active gastrointestinal symptoms or disease
* Prior gastrointestinal surgery that could interfere with conduct or interpretation of the studies (gastric bypass, gastric sleeves, esophagectomy, vagal nerve stimulators, etc)
* Pregnancy or breast-feeding
* History of neurodegenerative disorders (Parkinson's disease, multiple sclerosis, dementia, documented autonomic dysfunction, amyotrophic lateral sclerosis, etc)
* Vulnerable population (dementia, severe intellectual disability etc)
* Any condition or personal circumstance that, in the opinion of the investigator, renders the subject unlikely or unable to comply with the full study protocol which could interfere with the study assessments
* Allergy to eggs, allergy to soy, allergy to oats, or other study products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Gastric emptying T half | Baseline, 1 week
  Gastric emptying T half is measured using gastric emptying scintigraphy, which involves taking a meal with radioactive tracer and measuring the time it takes for 50% of the meal to leave the stomach. Results are reported in minutes.

SECONDARY OUTCOMES:
Proportion emptied using the standard egg diet | 2 hours, 4 hours
  The proportion emptied is reported as the percentage of the tracer remaining in the stomach at timepoints of 2 and 4 hours.
Proportion emptied using the vegan diet alternative | 2 hours, 4 hours
  The proportion emptied is reported as the percentage of the tracer remaining in the stomach at timepoints of 2 and 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No